CLINICAL TRIAL: NCT02838017
Title: Tissue Adhesive Compared to Sterile Strips After Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Tissue Adhesive vs. Sterile Strips After Cesarean Delivery
Acronym: TASC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on results of an interim analysis, the study was halted for futility
Sponsor: Endeavor Health (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Beth Plunkett, Clinical Associate Professor, Maternal & Fetal Medicine, Obstetrics & Gynecology, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EH16-095
Record Dates: First submitted 2016-07-12; First posted 2016-07-20 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Wound Complication; Complications; Cesarean Section
MeSH Terms: interventions — Tissue Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tissue Adhesive (Experimental): Tissue Adhesive will be placed over subcuticular suture closure.
  Interventions: Device: Tissue Adhesive
- Steri-Strips (Active Comparator): Sterile strips will be placed over subcuticular suture closure.
  Interventions: Device: Sterile strips

INTERVENTIONS:
Device: Tissue Adhesive
  Other Names: Dermabond; Dermaflex; 2-octyl cyanoacrylate
  Arms: Tissue Adhesive
Device: Sterile strips
  Other Names: Steri-Strips
  Arms: Steri-Strips

SUMMARY:
The goal of this project is to identify a strategy to reduce wound complications in women who undergo cesarean delivery by Pfannenstiel skin incision. Currently, many Pfannenstiel skin incisions are closed by subcuticular sutures followed by either placement of sterile strips or tissue A\adhesive. Either sterile strips or tissue adhesive can be placed over the wound as a covering but it is unclear which may reduce wound complication rates. The hypothesis of this study is that tissue adhesive will result in a reduction in wound complication rates when compared to sterile strips. Previously published studies in non-obstetric populations have identified tissue adhesive as a potential intervention to reduce wound complications. The eligible population for this study will include women at NorthShore University HealthSystem Evanston Hospital and University of Chicago Hospital who will undergo primary or repeat cesarean delivery via Pfannenstiel skin incision. Women in the study will be randomized to receive either sterile strips or tissue adhesive. The primary outcome to be evaluated will be a composite of wound complication which will include drainage, cellulitis, hematoma, seroma and/or wound separation (partial or complete). Secondary endpoints to be investigated include cosmetic outcome, patient satisfaction, cost comparison, and difference in operative times.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing Pfannenstiel Cesarean delivery

Exclusion Criteria:

* Inability to provide informed consent in English
* Planned use of staples for skin closure
* Unavailability of research personnel to accomplish consent and randomization at the time of cesarean

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2016-11; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Plunkett, MD, Principal Investigator — Endeavor Health; Lena Braginsky, MD, Study Director — Endeavor Health
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - NorthShore Evanston Hospital, Evanston, Illinois
  - NorthShore Highland Park Hospital, Highland Park, Illinois

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentiﬁcation, will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available immediately after publication with no end date.
Access Criteria: Investigators may request data by contacting lbraginsky@northshore.org

REFERENCES:
- [Background] Souza EC, Fitaroni RB, Januzelli DM, Macruz HM, Camacho JC, Souza MR. Use of 2-octyl cyanoacrylate for skin closure of sternal incisions in cardiac surgery: observations of microbial barrier effects. Curr Med Res Opin. 2008 Jan;24(1):151-5. doi: 10.1185/030079908x253807. PMID 18034920
- [Background] Mackeen AD, Packard RE, Ota E, Berghella V, Baxter JK. Timing of intravenous prophylactic antibiotics for preventing postpartum infectious morbidity in women undergoing cesarean delivery. Cochrane Database Syst Rev. 2014 Dec 5;2014(12):CD009516. doi: 10.1002/14651858.CD009516.pub2. PMID 25479008
- [Background] Noorani A, Rabey N, Walsh SR, Davies RJ. Systematic review and meta-analysis of preoperative antisepsis with chlorhexidine versus povidone-iodine in clean-contaminated surgery. Br J Surg. 2010 Nov;97(11):1614-20. doi: 10.1002/bjs.7214. PMID 20878942
- [Background] Stamilio DM, Scifres CM. Extreme obesity and postcesarean maternal complications. Obstet Gynecol. 2014 Aug;124(2 Pt 1):227-232. doi: 10.1097/AOG.0000000000000384. PMID 25004353
- [Background] Tipton AM, Cohen SA, Chelmow D. Wound infection in the obese pregnant woman. Semin Perinatol. 2011 Dec;35(6):345-9. doi: 10.1053/j.semperi.2011.05.020. PMID 22108085
- [Background] Buresch AM, Van Arsdale A, Ferzli M, Sahasrabudhe N, Sun M, Bernstein J, Bernstein PS, Ngai IM, Garry DJ. Comparison of Subcuticular Suture Type for Skin Closure After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2017 Sep;130(3):521-526. doi: 10.1097/AOG.0000000000002200. PMID 28796687
- [Background] Daykan Y, Sharon-Weiner M, Pasternak Y, Tzadikevitch-Geffen K, Markovitch O, Sukenik-Halevy R, Biron-Shental T. Skin closure at cesarean delivery, glue vs subcuticular sutures: a randomized controlled trial. Am J Obstet Gynecol. 2017 Apr;216(4):406.e1-406.e5. doi: 10.1016/j.ajog.2017.01.009. Epub 2017 Jan 30. PMID 28153666
- [Derived] Braginsky L, Javellana M, Cleveland E, Elue R, Wang C, Boyle D, Plunkett BA. Tissue Adhesive Compared With Sterile Strips After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2019 Aug;134(2):295-301. doi: 10.1097/AOG.0000000000003367. PMID 31306319

RESULTS

PARTICIPANT FLOW:
Groups:
- Tissue Adhesive: Tissue Adhesive will be placed over subcuticular suture closure.
  Tissue Adhesive
- Sterile Strips: Sterile strips will be placed over subcuticular suture closure.
  Sterile strips
Period: Overall Study
Arm/Group | Tissue Adhesive | Sterile Strips
Started | 252 | 252
Completed | 238 | 241
Not Completed | 14 | 11
Not completed — Lost to Follow-up | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Steri-Strips: Sterile strips will be placed over subcuticular suture closure.
  Sterile strips
- Total: Total of all reporting groups
Arm/Group | Tissue Adhesive | Steri-Strips | Total
Number analyzed (Participants) | 252 | 252 | 504
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [30.0 to 36.0] | 33.5 [29.0 to 36.0] | 34 [29.0 to 36.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252 | 252 | 504
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 28 | 58
  Not Hispanic or Latino | 191 | 204 | 395
  Unknown or Not Reported | 31 | 20 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 121 | 139 | 260
  Black or African American | 74 | 65 | 139
  Asian | 29 | 31 | 60
  Other | 31 | 20 | 51
Nulliparity [Count of Participants; unit: Participants] | 25 | 25 | 50
Prior cesarean delivery [Count of Participants; unit: Participants] | 144 | 140 | 284
Body mass index at delivery [Median (Inter-Quartile Range); unit: kg/m^2] | 32.9 [28.5 to 38.0] | 33.5 [29.0 to 38.2] | 33.3 [28.8 to 38.0]
Diabetes mellitus [Count of Participants; unit: Participants] | 30 | 44 | 74
Hypertensive disorders [Count of Participants; unit: Participants] | 54 | 57 | 111
Tobacco use [Count of Participants; unit: Participants] | 13 | 8 | 21
Immunocompromised [Count of Participants; unit: Participants] | 4 | 3 | 7
Cesarean delivery while in labor [Count of Participants; unit: Participants] | 64 | 56 | 120
Chorioamnionitis [Count of Participants; unit: Participants] | 11 | 10 | 21
Blood loss [Median (Inter-Quartile Range); unit: mL] | 700.0 [494.8 to 903.8] | 745.0 [525.0 to 994.0] | 700.0 [502.8 to 945.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Complication
Description: Wound drainage, Cellulitis, Abscess, Hematoma, Seroma or Separation
Time Frame: 6-8 weeks from cesarean delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Tissue Adhesive | Sterile Strips
Number analyzed (Participants) | 238 | 241
Participants | 18 | 19

2. Secondary Outcome: Number of Participants With Readmission for Wound Complication
Time Frame: Within 8 weeks from cesarean delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Tissue Adhesive | Sterile Strips
Number analyzed (Participants) | 238 | 241
Participants | 1 | 1

3. Secondary Outcome: Satisfaction With Cesarean Scar
Description: The investigators will be using a modified validated Patient Scar Assessment Scale (PSAS) which assessed scar-related pain, itchiness, color, stiffness, irregularity and overall satisfaction with the scar. Each item on the PSAS has a 10-point scale, with 10 indicating the highest symptom severity or lowest satisfaction. The median score for each item was compared between groups.
  Please see website in links section for more details on this assessment tool.
Time Frame: 6-8 weeks from cesarean delivery
Population: Completion of the modified Patient Scar Assessment Scale was accomplished in 203/252 (80.6%) of women in the tissue adhesive group and 203/252 (80.6%) of women in the sterile strips group.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tissue Adhesive | Sterile Strips
Number analyzed (Participants) | 203 | 203
score on a scale | 1 [1.0 to 3.0] | 2 [1.0 to 4.0]

4. Secondary Outcome: Number of Participants Who Required an Office or Emergency Department Visit for Wound Complication
Description: The investigators will review medical records to assess for ambulatory visits for wound complaints
Time Frame: Within 8 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Tissue Adhesive | Sterile Strips
Number analyzed (Participants) | 238 | 241
Participants | 16 | 18

5. Secondary Outcome: Operative Time
Description: The investigators will review operative records to assess operative time
Time Frame: At time of delivery
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | Tissue Adhesive | Sterile Strips
Number analyzed (Participants) | 238 | 241
min | 58.5 [48.0 to 70.3] | 60 [51 to 72]

6. Secondary Outcome: Number of Participants Requiring Antibiotic Treatment for Wound Complication
Description: The investigators will review medical records to assess for antibiotic prescriptions for wound complications
Time Frame: Within 8 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Tissue Adhesive | Sterile Strips
Number analyzed (Participants) | 238 | 241
Participants | 7 | 12

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Patients were contacted and medical records reviewed to assess for adverse events
Arm/Group | Tissue Adhesive | Sterile Strips
All-Cause Mortality (participants affected / at risk) | 0/252 | 0/252
Serious Adverse Events (participants affected / at risk) | 0/252 | 0/252
Other Adverse Events (participants affected / at risk) | 0/252 | 0/252

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT02838017/Prot_SAP_000.pdf